CLINICAL TRIAL: NCT03917602
Title: Human Amniotic Membrane Plug for Large Macular Holes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Mahmoud Abouhussein, Assistant professor, University of Alexandria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12042019
Record Dates: First submitted 2019-04-14; First posted 2019-04-17 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Macular Holes
Keywords: Human amniotic membrane; large macular holes
MeSH Terms: conditions — Retinal Perforations | interventions — Vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with large macular holes (Experimental): Patients suffering from large macular holes as documented by spectral domain OCT will undergo pars plan vitrectomy with human amniotic membrane insertion into the macular hole.
  Interventions: Procedure: human amniotic membrane plug with vitrectomy

INTERVENTIONS:
Procedure: human amniotic membrane plug with vitrectomy — using human amniotic membrane plug with vitrectomy to try to close large macular hole
  Other Names: human amniotic membrane plug with vitrectomy for closure of large macular holes

SUMMARY:
This is a prospective, interventional, consecutive case series conducted in Alexandria university. The aim of the study is to evaluate the therapeutic efficacy of human amniotic membrane in promoting closure of large macular holes.

DETAILED DESCRIPTION:
This is a prospective, interventional, consecutive case series conducted in Alexandria university. The aim of the study is to evaluate the therapeutic efficacy of human amniotic membrane in promoting closure of large macular holes.

Included participants with large macular holes will undergo complete vitrectomy is performed with an accurate vitreal base shaving (Constellation; Alcon Surgical). A human amniotic membrane hAM plug is taken from the hAM patch, and the final dimensions are adjusted with vitreoretinal scissors before insertion into the vitreous. The hAM plug is rolled inside the vitreoretinal forceps and inserted through the trocar into the vitreous. Then the human amniotic membrane is transplanted through macular hole into the subretinal space; it is then spread to cover the entire portion of the hole. Afterward, perfluorocarbon is injected to a complete overfilling of the break to permit good adhesion of the hAM plug to the underlying RPE and the overlying retina. Fluid-air exchange and an endotamponade injection is performed at the end of surgery.

ELIGIBILITY:
Inclusion Criteria:

* large macular hole confirmed by optical coherence tomography

Exclusion Criteria:

* patients who had diabetic retinopathy, vascular occlusion, retinal neovascularization, inflammatory disease and optic atrophy

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-05-11 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
closure of the macular hole | at the 6 month follow up visit
  closure of the macular hole as shown by optical coherence tomography

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
optical coherence tomography data of patients pre and postoperatively may be shared with other researchers
Supporting Information: Study Protocol
Time Frame: after start of recruiting patients